CLINICAL TRIAL: NCT03373045
Title: The CHRONICLE Study: A Longitudinal Prospective Observational Study of the Characteristics, Treatment Patterns and Health Outcomes of Individuals With Severe Asthma in the United States
Brief Title: Observational Study of Characteristics, Treatment and Outcomes With Severe Asthma in the United States (CHRONICLE)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry); MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00023
Record Dates: First submitted 2017-11-20; First posted 2017-12-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: Severe asthma; Monoclonal antibody; Corticosteroid; Non-interventional
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of US adults with severe asthma: To describe patient characteristics, treatment patterns, and health outcomes among a large, geographically diverse cohort of US adults with severe asthma who are not controlled on high-dose ICS with additional controllers and/or require chronic systemic corticosteroid or monoclonal antibody therapy.

SUMMARY:
The CHRONICLE Study is a multi-center, non-interventional, prospective cohort study of adults with severe asthma who do not achieve control with high-dose inhaled corticosteroid (ICS) therapy with additional controllers and/or require systemic corticosteroid or monoclonal antibody therapy. Data will be collected from the healthcare provider in a uniform manner for every patient enrolled using an electronic case report form (eCRF). Data will be collected monthly from patients via web-based surveys. Patients will be followed until study discontinuation or the patient withdraws from the study or death, whichever occurs first. The expectation is that patients will be followed for a period of at least 3 years.

DETAILED DESCRIPTION:
The CHRONICLE Study is a multi-center, non-interventional, prospective cohort study of adults with severe asthma who do not achieve control with high-dose ICS therapy with additional controllers and/or require systemic corticosteroid or monoclonal antibody therapy. This study will provide a contemporary description of the epidemiology and medical management of United States adults with severe asthma who have not achieved control with high-dose ICS therapy and additional controllers. Additionally, the study will describe the use of and outcomes associated with recently approved monoclonal antibody therapies for severe asthma. Patients will be enrolled from a diverse population of academic and community-based specialist centers across the US. Data will be collected in a naturalistic manner and patient management will not be influenced by the study protocol. At least 1500 patients in the US with a confirmed diagnosis of severe asthma will be enrolled by a diverse set of asthma specialists (eg, allergists and pulmonologists who treat asthma) from academic and community-based centers. Basic de-identified information will be collected for all patients meeting study inclusion criteria, including those not approached for enrollment or who decline enrollment, to enable an assessment of the enrolled and non-enrolled populations. This information will include age, sex, insurance status, age at asthma diagnosis, class of asthma treatment per study inclusion criteria, number of asthma exacerbations in the past 12 months, study eligibility, whether the patient was approached for enrollment, study enrollment status, and reason for not enrolling for those who are approached but do not enroll. Patient-reported asthma control (Asthma Control Test [ACT]), asthma exacerbations, and treatment adherence will be solicited monthly. Patient-reported information on asthma-related healthcare utilization, global evaluation of treatment effectiveness (GETE), and work productivity (Work Productivity and Activity Impairment Asthma questionnaire [WPAI-Asthma]) will be collected at baseline and approximately every 3 months. Detailed information on asthma-related quality of life (Saint George's Respiratory Questionnaire [SGRQ]) as well as presence of an asthma treatment plan will be collected from patients approximately every 6 months. All of the questionnaires will be collected via web-based surveys. Patients will then be followed until study discontinuation or the patient withdraws from the study or death, whichever occurs first. The expectation is that patients will be followed for a period of at least 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a diagnosis of severe asthma for at least 12 months prior to enrollment and confirmed by the Investigator not to be due to alternative diagnoses.

2. Currently receiving care from specialist physicians (eg, pulmonologists and or allergists) at the Investigator's or sub-investigator's site.

3. 18 years of age and older. 4. Meeting at least one of the following three criteria (a, b, or c):

a. Uncontrolled asthma while receiving high-dose ICS with additional controllers.

i. Uncontrolled is defined by meeting at least one of the following (as outlined by ATS/ERS [American Thoracic Society/European Respiratory Society] guidelines):

1. Poor symptom control: Asthma Control Questionnaire consistently ≥1.5, ACT <20 (or "not well controlled" by NAEPP [National Asthma Education and Prevention Program]/Global Initiative for Asthma guidelines).
2. Frequent severe exacerbations: two or more bursts of systemic corticosteroids (≥3 days each) in the previous 12 months.
3. Serious exacerbations: at least one hospitalization, intensive care unit stay or mechanical ventilation in the previous 12 months.
4. Airflow limitation: after appropriate bronchodilator withhold FEV1 <80% predicted (in the face of reduced FEV1/FVC defined as less than the lower limit of normal).

ii. For the purposes of this study, high-dose ICS will be defined as

1. ICS at a cumulative dose of >500 μg fluticasone propionate equivalents daily as defined in Appendix A, or 2. Highest labeled dose of a combination of ICS/LABA. b. Current use of a Food and Drug Administration (FDA)-approved monoclonal antibody agent for treatment of severe asthma (use is not primarily for an alternative condition).

c. Use of systemic corticosteroids or other systemic immunosuppressants (any dose level) for approximately 50% or more of the prior 12 months for treatment of severe asthma (use is not primarily for an alternative condition).

Exclusion Criteria

1. Not willing and able to sign written informed consent. Consent can be obtained from having a responsible, legally authorized representative acting on patient's behalf.
2. Not fluent in English or Spanish.
3. Inability to complete study follow-up or web-based PROs. If the patient does not have email or web access, minimal assistance from others to access the web-based PRO is permitted (ie receiving the email and/or assisting patient in navigating to the web page); PROs must be completed by the patient.
4. Received an investigational therapy for asthma, allergy, atopic disease, or eosinophilic disease as part of a clinical trial during the 6 months prior to enrollment.

   1. Once enrolled in the CHRONICLE Study, patients can enroll in trials of investigational therapies (as well as other non-interventional studies) as long as they continue to complete study follow-up. If a patient enrolls in a trial of an investigational therapy, the identity (National Clinical Trial [NCT] number) of the study and dates of the first and last investigational therapy administrations will be collected. If a patient receives blinded therapy in a trial, the Investigator will request the identity of that therapy at trial conclusion so that treatment information collected for the current study may be updated accordingly.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is estimated that at least 1500 patients in the US with a confirmed diagnosis of severe asthma will be enrolled by a diverse set of asthma specialists (eg, allergists and pulmonologists who treat asthma) from academic and community-based centers.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization- hospitalizations, clinic Visits, and asthma exacerbations | At baseline, every 6 months, through study completion, assessed up to 7 years.
  Longitudinal changes of Healthcare utilization will be measured using directly collected information from medical, hospital, and pharmacy records to provide a supplementary comprehensive assessment of each patient's healthcare utilization during the study period.
Asthma treatment | At baseline, every 6 months, through study completion, assessed up to 7 years.
  Asthma medications with dose and start/stop dates including all FDA-approved and standard of care treatments for asthma will be assessed. Longitudinal changes in asthma treatment will also be assessed.
Treatment adherence | At baseline, every 1 month, through study completion, assessed up to 7 years.
  Extraction of electronic medical, hospital, and pharmacy records will take place at study close and potentially at interim time points to provide a supplementary assessment of each patient's healthcare resource utilization. Longitudinal changes in patient reported treatment adherence will also be assessed.
Asthma control test (ACT) | Change from baseline, every 1 month, through study completion, assessed up to 4 years.
  Patient-reported asthma symptoms and control will be collected via the ACT questionnaire; a 5 item, self-administered survey that is designed to help the patient describe their asthma and how it affects their daily activities. ACT questionnaire is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).
  In 2022, the ACT survey will be removed, and only the AIRQ will be solicited monthly.
Patient-reported asthma exacerbations | Change from baseline, every 1 month, through study completion, assessed up to 4 years.
  Asthma exacerbations, the primary analytical definition will be worsening of asthma that leads to any of the following: Use of systemic corticosteroids (or a temporary increase in a stable corticosteroid background dose) for at least 3 days; a single depo-injectable dose of corticosteroids will be considered equivalent to a 3-day course of systemic corticosteroids. An emergency department or urgent care visit (defined as evaluation and treatment for <24 hours in an emergency department or urgent care center) due to asthma that required systemic corticosteroids. An inpatient hospitalization (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥24 hours) due to asthma.
  In 2022, the asthma exacerbations survey will be removed, and only the AIRQ will be solicited monthly.
Asthma Impairment and Risk Questionnaire (AIRQ) | At baseline, every 1 month, through study completion, assessed up to 4 years
  AIRQ is a 10-item, equally weighted, yes/no composite asthma control questionnaire that includes 7 impairment and 3 risk items. AIRQ scores range from 0 to 10, with lower scores representing better controlled asthma.
Work Productivity and Activity Impairment Asthma questionnaire (WPAI-Asthma) | At baseline, every 3 months, through study completion, assessed up to 7 years.
  Patient-reported productivity impairment assessment including work productivity, activity impairment, and disability will be collected via the WPAI-Asthma. Information will only be collected from procedures that are part of the patient's routine clinical care. WPAI Asthma questionnaire is calculated from 0 to 10 score (0 indicates-Asthma had no effect on my work/ daily activities and 10 indicates Asthma completely prevented me from working score/ doing my daily activities).
St. George's Respiratory Questionnaire (SGRQ) | At baseline, every 6 months, through study completion, assessed up to 7 years.
  Patient-reported assessment of asthma quality of life will be collected via the SGRQ. SGRQ, a disease specific health-related quality of life measure developed for both asthma and chronic obstructive pulmonary disease (COPD) patients. The SGRQ has 50 items and scores are calculated for 3 domains (symptoms, activity, and impact [psychosocial]) as well as total score.
  Symptoms - this component is concerned with the effect of respiratory symptoms, their frequency and severity.
  Impacts (psychosocial) - covers a range of aspects concerned with social functioning and psychological disturbances resulting from respiratory disease Activity - concerned with activities that cause or are limited by breathlessness. Total score summarizes the impact of the disease on overall health status.
  The score is expressed as a percentage of overall impairment, where 100 represents worst possible health status and 0 indicates best possible health status.
Global evaluation of treatment effectiveness (GETE) | At baseline, every 6 months, through study completion, assessed maximum up to 7 years.
  Patient evaluation of asthma treatment effectiveness will be measured using GETE; a simple measure of perceived treatment effectiveness. The patient will grade the overall treatment effectiveness using the following criteria: excellent (complete control of asthma); good (marked improvement of asthma); moderate (discernible, but limited improvement in asthma); poor (no appreciable change in asthma); or worsening (of asthma).
Number of Participants With Adverse Events associated with corticosteroid therapy | At baseline, every 6 months, through study completion, assessed up to 7 years.
  Frequency of relevant medical events such as weight gain (change in BMI), hypertension, dyslipidemia, pneumonia, bone densitometry results, osteoporosis / osteopenia, hip and spinal fractures, avascular necrosis, cataract, glaucoma, diabetes mellitus, cardiovascular disease, Cushing's syndrome, adrenal insufficiency, peptic ulcer disease, myopathy, pseudotumor cerebri, mood disturbance, and insomnia or sleep disturbance.
Relevant respiratory medical events | At baseline, every 6 months, through study completion,assessed up to 7 years.
  Frequency of relevant respiratory medical events such as pneumonia, pleural effusion, chronic bronchitis, allergic rhinitis.
Respiratory comorbidities | At baseline, every 6 months, through study completion, assessed up to 7 years.
  Prevalence of respiratory comorbidities such as chronic obstructive pulmonary disease (COPD), bronchiectasis, alpha-1 anti-trypsin deficiency, Churg- Strauss syndrome (eosinophilic granulomatosis with polyangiitis [EGPA]), airway stenosis, cystic fibrosis, allergic bronchopulmonary aspergillosis,chronic eosinophilic pneumonia, bronchiolitis obliterans, immunodeficiency, primary ciliary dyskinesia, atelectasis, arterial hypertension, pulmonary hypertension, neuromuscular disease, allergic rhinitis, chronic rhinosinusitis, and pulmonary embolism.
Non-respiratory comorbidities | At baseline, every 6 months, through study completion, assessed up to 7 years.
  Prevalence of non-respiratory comorbidities such as diabetes, thyroid disease, cardiac disease, etc.
Events of special interest | At baseline, every 6 months, through study completion, assessed up to 7 years.
  Frequency of special interest events including new onset malignancy, severe infection, anaphylaxis, or mortality.
Complete blood count with differential including blood eosinophil count. | Change from baseline, every 6 months, through study completion, assessed up to 7 years.
  To assess complete blood count with differential including blood eosinophil count as a variable for asthma evaluation.
Total immunoglobulin E (IgE) | Change from baseline, every 6 months, through study completion, assessed up to 7 years.
  To assess total IgE as a variable for asthma evaluation.
Radiographic changes in asthma evaluation. | Change from baseline, every 6 months, through study completion, assessed up to 7 years.
  Radiographic changes in asthma evaluation included chest X-rays (dates, views, description of major chest findings), Chest computed tomography scan (dates, high resolution (yes/no), intravenous contrast (yes/no), description of major findings). Radiographic asthma evaluation conducted as part of routine care.
Forced Vital Capacity (FVC) | Change from baseline, every 6 months, through study completion, assessed up to 7 years.
  FEV1 (liters and % predicted) will be assessed as a variable for asthma evaluation.
Forced Expiratory Volume in 1 second (FEV1) | Change from baseline, every 6 months, through study completion, assessed up to 7 years.
  FEV1 (liters and % predicted) will be assessed as a variable for asthma evaluation.
Fractional exhaled nitric oxide (FENO) | Change from baseline, every 6 months, through study completion, assessed up to 7 years.
  To assess FENO as a variable for asthma evaluation.

CONTACTS AND LOCATIONS:
Locations (150):
- United States (149):
  - Research Site, Birmingham, Alabama
  - Research Site, Hoover, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Modesto, California
  - Research Site, Redondo Beach, California
  - Research Site, Riverside, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Studio City, California
  - Research Site, Ventura, California
  - Research Site, Westminster, California
  - Research Site, Aurora, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Farmington, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lake Mary, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Plantation, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Albany, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Villa Rica, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Glen Ellyn, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Georgetown, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Rockville, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Burlington, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Clinton Township, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Hamtramck, Michigan
  - Research Site, Wyoming, Michigan
  - Research Site, Maplewood, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Plymouth, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Brick, New Jersey
  - Research Site, Marlton, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, North Bergen, New Jersey
  - Research Site, Northfield, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Bayside, New York
  - Research Site, Brooklyn, New York
  - Research Site, Corning, New York
  - Research Site, Great Neck, New York
  - Research Site, Jamaica, New York
  - Research Site, Mineola, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New Paltz, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Rockville Centre, New York
  - Research Site, Staten Island, New York
  - Research Site, The Bronx, New York
  - Research Site, Valhalla, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Corvallis, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Blue Bell, Pennsylvania
  - Research Site, DuBois, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Clinton, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Aransas Pass, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Dallas, Texas
  - Research Site, Denison, Texas
  - Research Site, Duncanville, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Live Oak, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Murray, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Lynchburg, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Vancouver, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Greenfield, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Onalaska, Wisconsin
  - Research Site, Wausau, Wisconsin
- Research Site, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Panettieri RA Jr, Mohan A, Lugogo NL, Ledford DK, Carstens DD, Ambrose CS. Outcomes after biologic initiation among patients with severe asthma and normal lung function in the CHRONICLE study. Respir Res. 2026 Jan 7;27(1):5. doi: 10.1186/s12931-025-03439-8. PMID 41501790
- [Derived] Ledford DK, Carr WW, Moore WC, Lugogo NL, Mohan A, Chipps B, Mackie AR, Lindsley AW, Spahn J, Ambrose CS. Reduced Effectiveness of Anti-IgE Treatment Among Adults with Severe Asthma with Older Age of Asthma Onset: Results from the CHRONICLE Study. J Asthma Allergy. 2024 Oct 9;17:977-982. doi: 10.2147/JAA.S476774. eCollection 2024. PMID 39398317
- [Derived] Ledford DK, Soong W, Carr W, Trevor J, Tan L, Carstens D, Ambrose CS. Real-world severe asthma biologic administration and adherence differs by biologic: CHRONICLE study results. Ann Allergy Asthma Immunol. 2023 Nov;131(5):598-605.e3. doi: 10.1016/j.anai.2023.07.017. Epub 2023 Jul 26. PMID 37506846
- [Derived] Chipps BE, Soong W, Panettieri RA Jr, Carr W, Gandhi H, Zhou W, Cook B, Llanos JP, Ambrose CS. Number of patient-reported asthma triggers predicts uncontrolled disease among specialist-treated patients with severe asthma. Ann Allergy Asthma Immunol. 2023 Jun;130(6):784-790.e5. doi: 10.1016/j.anai.2023.03.001. Epub 2023 Mar 10. PMID 36906262
- [Derived] Panettieri RA Jr, Ledford DK, Chipps BE, Soong W, Lugogo N, Carr W, Mohan A, Carstens D, Genofre E, Trudo F, Ambrose CS. Biologic use and outcomes among adults with severe asthma treated by US subspecialists. Ann Allergy Asthma Immunol. 2022 Oct;129(4):467-474.e3. doi: 10.1016/j.anai.2022.06.012. Epub 2022 Jun 19. PMID 35728746
- [Derived] Panettieri RA Jr, Chipps BE, Moore WC, Soong W, Carr WW, Kreindler JL, O'Quinn S, Trudo F, Ambrose CS. Differing perceptions of asthma control and treatment effectiveness by patients with severe asthma and treating subspecialists in the United States. J Asthma. 2022 Sep;59(9):1859-1868. doi: 10.1080/02770903.2021.1963766. Epub 2021 Nov 5. PMID 34374622
- [Derived] Trevor J, Lugogo N, Carr W, Moore WC, Soong W, Panettieri RA Jr,, Desai P, Trudo F, Ambrose CS. Severe asthma exacerbations in the United States:: Incidence, characteristics, predictors, and effects of biologic treatments. Ann Allergy Asthma Immunol. 2021 Nov;127(5):579-587.e1. doi: 10.1016/j.anai.2021.07.010. Epub 2021 Jul 15. PMID 34273485
- [Derived] Soong W, Chipps BE, O'Quinn S, Trevor J, Carr WW, Belton L, Trudo F, Ambrose CS. Health-Related Quality of Life and Productivity Among US Patients with Severe Asthma. J Asthma Allergy. 2021 Jun 25;14:713-725. doi: 10.2147/JAA.S305513. eCollection 2021. PMID 34211280
- [Derived] Ambrose CS, Chipps BE, Moore WC, Soong W, Trevor J, Ledford DK, Carr WW, Lugogo N, Trudo F, Tran TN, Panettieri RA Jr. The CHRONICLE Study of US Adults with Subspecialist-Treated Severe Asthma: Objectives, Design, and Initial Results. Pragmat Obs Res. 2020 Jul 16;11:77-90. doi: 10.2147/POR.S251120. eCollection 2020. PMID 32765156
- [Derived] Moore WC, Panettieri RA Jr, Trevor J, Ledford DK, Lugogo N, Soong W, Chipps BE, Carr W, Belton L, Gandhi H, Trudo F, Ambrose CS. Biologic and maintenance systemic corticosteroid therapy among US subspecialist-treated patients with severe asthma. Ann Allergy Asthma Immunol. 2020 Sep;125(3):294-303.e1. doi: 10.1016/j.anai.2020.04.004. Epub 2020 Apr 15. PMID 32304877
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00023&attachmentIdentifier=392eea35-d61a-43f9-83a7-da2675002f5b&fileName=D3250R00023_CSR_Synopsis.pdf&versionIdentifier=